CLINICAL TRIAL: NCT06838806
Title: Differentiating Benign and Malignant Pulmonary Nodules Using Epigenetically Modified Nucleosomes in Plasma
Brief Title: Epigenetic Nucleosomes in Plasma for Pulmonary Nodule Differentiation
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Volition Diagnostics UK Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202412107RIND
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Lung Nodule
Keywords: liquid biopsy; epigenetic
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — whole blood into a K2 EDTA tube and whole blood into a cell-free DNA BCT tube.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood draw — Plasma samples will be collected in NTU Hospital or NTUCC. ChLIA kits and all other reagents will be provided by Volition. ChLIA analysis of samples will be performed by a Volition designated laboratory in Taiwan( NTU Centres of Genomic and Precision Medicine).

SUMMARY:
Investigators aim to evaluate the diagnostic accuracy of the Nu.Q blood test for lung cancer in the Taiwanese population and compare its diagnostic performance with low-dose computed tomography (LDCT) or computed tomography (CT). Additionally, investigators will investigate the potential role of Nu.Q in lung cancer prevention and its impact on survival outcomes.

Study Method:

Investigators plan to collect 20 mL of blood samples from individuals undergoing chest LDCT/CT, isolate plasma for Nu.Q™ analysis, and compare the results with corresponding lung cancer pathology findings. The estimated sample size is 500 participants.

DETAILED DESCRIPTION:
Currently, early lung cancer screening primarily relies on low-dose computed tomography (LDCT) of the chest. However, blood tests offer a more convenient alternative. Despite this, existing blood tests lack sufficient accuracy and sensitivity for lung cancer screening. Developing a reliable blood-based screening tool could significantly enhance the detection rate and accuracy of early lung cancer screening.

Previous studies have shown that nucleosomes undergo variations during early cancer development. The Belgian company Volition has developed a blood test method based on chemiluminescence immunoassay (ChLIA) to measure nucleosomes in the blood, branded as Nu.Q™. Preliminary studies have demonstrated that Nu.Q™ can detect abnormal nucleosome biomarkers associated with early lung cancer.

This study, in collaboration with Volition, will collect 20 mL of blood samples from individuals undergoing chest LDCT. Plasma will be isolated and analyzed using Nu.Q™ at the National Taiwan University Center for Genomics and Precision Medicine. The test results will be compared with corresponding lung cancer medical records, LDCT findings, and pathological diagnoses. The study aims to enroll 500 participants.

The objectives of this study are to validate the diagnostic accuracy of the Nu.Q™ blood test for lung cancer in the Taiwanese population, compare its diagnostic performance with LDCT, and explore its potential role in lung cancer prevention and improved survival outcomes. This study is conducted as an industry-academic collaboration project with National Taiwan University.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 or older
* Underwent a low-dose chest CT scan or a standard chest CT scan, showing lung nodules ≥ 6mm
* Individuals understand the content of the consent form and are willing to participate in this study.
* The lung nodule is assessed by a physician as high-risk, requiring thoracic surgery or biopsy for diagnosis

Exclusion Criteria:

* Pregnant women
* Individuals without capacity for consent, unable to understand the content of the consent form, or unwilling to participate in this study
* Assessed by a physician as unsuitable for thoracic surgery or biopsy for diagnosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study would involve collection of plasma samples with informed consent from 500 people who already receive a chest tomography or low dose chest tomography.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The endpoint is pathology result of diagnosis. | 2 weeks
  pathology result according to the formal pathology report.

SECONDARY OUTCOMES:
long-term cancer related outcomes | 4 years
  The long-term outcomes will include occurrence of Lung cancer, cancer related death and overall death.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No